CLINICAL TRIAL: NCT03239080
Title: Effect of RANKL Inhibition on Healing of Bone Erosion in Rheumatoid Arthritis Using HR-pQCT
Brief Title: Effect of Denosumab in Erosion Healing in RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA-RANKL-2017
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; HR-pQCT; erosion; denosumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Denosumab (Active Comparator): Subcutaneous injections of denosumab 60mg will be given in 4 doses at each visit (at baseline, 6, 12 and 18 months).
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): Subcutaneous injections of placebo (0.9% Sodium Chloride solution) will be given in 4 doses at each visit (at baseline, 6, 12 and 18 months).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Denosumab — Subcutaneous injections of denosumab 60mg will be given in 4 doses at each visit (at baseline, 6, 12 and 18 months).
  Arms: Denosumab
Other: Placebo — Subcutaneous injections of placebo (0.9% Sodium Chloride solution) will be given in 4 doses at each visit (at baseline, 6, 12 and 18 months).
  Arms: Placebo

SUMMARY:
To evaluate the effects of denosumab on erosion healing and change in physical function in RA patients.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study, which aimed to evaluate the effects of denosumab on erosion healing and change in physical function in rheumatoid arthritis (RA) patients in low-disease activity or remission receiving synthetic DMARDs (sDMARDs) treatment using High-resolution peripheral quantitative CT (HR-pQCT).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* DAS28 ≤5.1
* without severe deformity in MCP joints which would influence the longitudinal assessment of HR-pQCT

Exclusion Criteria:

* RA functional status class IV (limited in ability to perform usual self-care, vocational, and avocational activities)
* treatment with any biologic DMARDs for RA treatment within 8 weeks before randomisation
* pregnancy or premenopausal women planning pregnancy
* previous use of denosumab, zoledronic acid or teriparatide
* Hyperparathyroidism
* contraindications to denosumab
* Bisphosphonate, biologic DMARDs and the use of oral glucocorticoid >10 mg/day (prednisolone equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with erosion healing determined using HR-pQCT on MCP 2-4 | 12 months
  1). A decrease in erosion volume of ≥ smallest detectable change (SDC) from baseline, and 2). The presence of > SDC in osteosclerosis at the margin of erosion.
The percentage of patients with erosion healing determined using HR-pQCT on MCP 2-4 | 24 months
  1). A decrease in erosion volume of ≥ smallest detectable change (SDC) from baseline, and 2). The presence of > SDC in osteosclerosis at the margin of erosion.

SECONDARY OUTCOMES:
Erosion progression | 12 and 24 month
  Changes in size of erosion (depth, width and volume) and marginal osteosclerosis (semi-quantitative and quantitative) using HR-pQCT
Radiographic progression | 12 and 24 months
  Radiographic progression expressed by changes in van der Heijde-Sharp score on radiograph
Change in various patient-reported outcomes | 12 and 24 month
  Changes in physical function (HAQ) will be measured
Association between the changes in erosion size on HR-pQCT, van der Heijde-Sharp score on radiograph and HAQ | 24 month
  Association between the changes in erosion size on HR-pQCT, van der Heijde-Sharp score on radiograph and HAQ will be analysed
Changes in joint space width (minimal, maximal, asymmetry and distribution) using HR-pQCT | 12 and 24 month
  Changes in joint space width (minimal, maximal, asymmetry and distribution) using HR-pQCT

CONTACTS AND LOCATIONS:
Overall Officials: Lai Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine and Therapeutics, Hong Kong, China

REFERENCES:
- [Derived] So H, Cheng IT, Lau SL, Chow E, Lam T, Hung VW, Li EK, Griffith JF, Lee VW, Shi L, Huang J, Kwok KY, Yim CW, Li TK, Lo V, Lee J, Lee JJ, Qin L, Tam LS. Effects of RANKL inhibition on promoting healing of bone erosion in rheumatoid arthritis using HR-pQCT: a 2-year, randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2021 Aug;80(8):981-988. doi: 10.1136/annrheumdis-2021-219846. Epub 2021 Apr 2. PMID 33811034